CLINICAL TRIAL: NCT05460832
Title: A Randomised, Double-Blind, Placebo-Controlled, Dose-Ranging Phase 2b Study to Investigate the Efficacy & Safety of MBS2320 in Participants With Moderate to Severe Active Rheumatoid Arthritis With Inadequate Response to Methotrexate Alone
Brief Title: Phase 2b Study of MBS2320 in Participants With Methotrexate-Refractory RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Modern Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IST-06; 2020-005496-13 (EudraCT Number)
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis (RA); MBS2320
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MBS2320 5 mg (Experimental)
  Interventions: Drug: MBS2320 5 mg
- MBS2320 20 mg (Experimental)
  Interventions: Drug: MBS2320 20 mg
- MBS2320 40 mg (Experimental)
  Interventions: Drug: MBS2320 40 mg

INTERVENTIONS:
Drug: MBS2320 5 mg — Oral capsule
  Arms: MBS2320 5 mg
Drug: MBS2320 20 mg — Oral capsule
  Arms: MBS2320 20 mg
Drug: MBS2320 40 mg — Oral capsule
  Arms: MBS2320 40 mg
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis (RA) affects 1 percent of the population worldwide and up to 40 percent of patients don't respond to current treatments. MBS2320, the drug being tested in this trial, represents a new approach to treating RA, with the potential not only to reduce levels of inflammation but to also directly prevent bone damage. The aim of this project is to test the safety, tolerability and efficacy of MBS2320 in patients with RA in combination with an existing treatment, methotrexate.

Approximately 224 participants with moderate to severe active RA who have not responded to treatment with Methotrexate will be enrolled from around 45 to 55 sites around the world. Participants will be randomly assigned to receive 1 of 3 doses of MBS2320 (5 mg, 20 mg, or 40 mg) or placebo (a "dummy" drug).

The maximum duration of study participation for a participant will be 22 weeks, which consists of a Screening Period of up to 4 weeks, Treatment Period of 12 weeks, and a Follow-up Period of 6 weeks.

Participants on the study will be asked to attend the hospital or clinic for regular visits during which they will have planned study assessments to evaluate the effectiveness, tolerability and safety of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with RA based on either the 1987-revised ACR classification criteria or the 2010 ACR/ EULAR criteria for ≥3 months prior to screening.
2. Has active RA as defined by the following minimum disease activity criteria:

   * ≥6 swollen joints (based on 66 joint counts)
   * ≥6 tender joints (based on 68 joint counts)
   * hsCRP > upper limit of normal reference range (ULN)
3. Considered to be inadequately responding to oral or parenteral MTX therapy for ≥3 months and <10 years prior to screening and to be tolerating a dose of 15 to 25 mg per week. Participants should also be on a stable dose of folic acid (or equivalent).
4. Except for MTX, must have discontinued all oral DMARDs prior to baseline visit.
5. If participants are taking NSAIDs or acetaminophen for stable medical conditions, they should be receiving these medications at a stable dose for at least 4 weeks prior to baseline visit and the doses of the medications should be kept stable throughout the study.
6. If participants are taking oral corticosteroids (equivalent to prednisolone ≤10 mg), or inhaled corticosteroids, they should be receiving these medications at a stable dose for at least 4 weeks prior to baseline visit for stable medical conditions.

This list contains only key inclusion criteria.

Exclusion Criteria:

1. Abnormality in the 12-lead ECG, heart rate or blood pressure at screening.
2. Any clinically significant neurological, GI, renal, hepatic, CV, psychiatric, respiratory, metabolic, endocrine, haematological, ophthalmic, or other major disorder which, in the opinion of the Investigator, would put the participant at risk by participating in the study.
3. Any current malignancy or a history of malignancy within 5 years prior to screening, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
4. Any other inflammatory or arthritic disease in addition to RA that may interfere with the study.
5. Active infection that is clinically significant in the Investigator's opinion, or any infection requiring hospitalisation or treatment with intravenous antimicrobials ≤60 days of screening, or any infection requiring oral antimicrobial therapy ≤2 weeks of the baseline visit.
6. Clinically significant features of arthroses that could interfer with study assessments and objectives.

This list contains only key exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: IST-06 IST-06, Study Director — Modern Biosciences Ltd
Locations (46):
- Bosnia and Herzegovina (3):
  - Site 1201 - Univerzitetski Klinicki Centar Republike Srpske, Banja Luka
  - Site 1204 - Univerzitetski Klinicki Centar Republike Srpske, Banja Luka
  - Site 1202 - General Hospital Gradiška, Gradiška
- Bulgaria (7):
  - Site 1308 - Medical Center Medconsult Pleven OOD, Pleven
  - Site 1302 - Medical Center Artmed OOD, Plovdiv
  - Site 1303 - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - Site 1306 - Diagnostic- Consultative Center Convex EOOD, Sofia
  - Site 1307 - Medical Center Excelsior OOD - PPDS, Sofia
  - Site 1301 - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
  - Site 1304 - Medical Center Leo Clinic EOOD, Varna, Varna
- Chile (7):
  - Site 2103 - Enroll SpA - PPDS, Providencia
  - Site 2105 - CTR Estudios, Providencia
  - Site 2104 - Meditek Ltda, Santiago
  - Site 2106 - Biocinetic SpA, Santiago
  - Site 2107 - Hospital Dr Sotero Del Rio, Santiago
  - Site 2102 - Clinical Research Chile SpA - PPDS, Valdivia
  - Site 2101 - Oncocentro APYS, Viña del Mar
- Czechia (4):
  - Site 1104 - CCR Ostrava s.r.o., Ostrava
  - Site 1101 - CCR Czech, Pardubice
  - Site 1103 - CLINTRIAL s.r.o., Prague
  - Site 1102 - MEDICAL PLUS, s.r.o., Uherské Hradište
- Guatemala (5):
  - Site 2401 - Clinica Medica Con Especialidad Reumatologia, Guatemala City
  - Site 2402 - Clinica Medica Especializada en Reumatologia, Guatemala City
  - Site 2404 - Reumacentro, Guatemala City
  - Site 2405 - Hospital Herrera Llerandi, Guatemala City
  - Site 2406 - Clinica Medica Especializada en Medicina Interna, Guatemala City
- Mexico (6):
  - Site 2206 - Centro de Alta Especialidad En Reumatologia E Investigacion Del Potosi SC, Burócratas del Estado
  - Site 2203 - Centro de Estudios de Investigacion Basica Y Clinica SC, Guadalajara
  - Site 2202 - Morales Vargas Centro de Investigacion SC, León
  - Site 2201 - Centro de Investigación en Artritis y Osteoporosis - PPDS, Mexicali
  - Site 2205 - Biológicos Especializados S.A. de C.V., Mexico City
  - Site 2204 - Centro de Investigación y Tratamiento Reumatológico S.C, Miguel Hidalgo
- Poland (8):
  - Site 1006 - ClinicMed Daniluk, Nowak Spółka Jawna, Bialystok
  - Site 1002 - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Site 1009 - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Site 1007 - NZOZ Lecznica MAK-MED, Nadarzyn
  - Site 1004 -Twoja Przychodnia NCM, Nowa Sól
  - Site 1001 - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Site 1003 - Centrum Medyczne Reuma Park NZOZ, Warsaw
  - Site 1008 - Centrum Medyczne AMED, Warsaw
- Serbia (6):
  - Site 1402 - Institute of Rheumatology Belgrade - PPDS, Belgrade
  - Site 1403 - Institute of Rheumatology Belgrade - PPDS, Belgrade
  - Site 1404 - Military Medical Academy, Belgrade
  - Site 1405 - Institute of Rheumatology Belgrade - PPDS, Belgrade
  - Site 1406 - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Site 1401 - Special Hospital For Rheumatic Diseases Novi Sad, Novi Sad

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MBS2320 5 mg | MBS2320 20 mg | MBS2320 40 mg
Started | 62 | 62 | 63 | 61
Completed | 57 | 61 | 54 | 57
Not Completed | 5 | 1 | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- MBS2320 5 mg: MBS2320 5 mg once daily for 12 weeks
- MBS2320 20 mg: MBS2320 20 mg once daily for 12 weeks
- MBS2320 40 mg: MBS2320 40 mg once daily for 12 weeks
- Placebo: Matching placebo capsules were provided containing the same excipients as the MBS2320 capsules but minus the active drug. The dosing instructions were the same as for MBS2320.
- Total: Total of all reporting groups
Arm/Group | MBS2320 5 mg | MBS2320 20 mg | MBS2320 40 mg | Placebo | Total
Number analyzed (Participants) | 62 | 63 | 61 | 62 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 54 | 54 | 52 | 209
  >=65 years | 13 | 9 | 7 | 10 | 39
Age, Continuous [Median (Standard Deviation); unit: Years] | 54.0 (13.82) | 55.0 (12.48) | 53.0 (11.26) | 55.5 (11.42) | 55.0 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 59 | 54 | 48 | 213
  Male | 10 | 4 | 7 | 14 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 11 | 11 | 5 | 39
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 39 | 45 | 39 | 47 | 170
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 7 | 11 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Successful Composite Clinical Response According to the Criteria for American College of Rheumatology 20% Response (ACR20)
Description: Achieving clinical response according to the criteria for ACR20:
  * ≥20% improvement in 68-Tender Joint Count;
  * ≥20% improvement in 66-SJC; and
  * ≥20% improvement in at least 3 of the 5 following parameters:
    1. Physician's global assessment of disease activity
    2. Participant's global assessment of disease activity
    3. Participant's assessment of arthritis pain
    4. Health Assessment Questionnaire - Disability Index (HAQ-DI)
    5. High-sensitivity C-reactive protein (hsCRP)
Time Frame: Week 12
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | MBS2320 5 mg | MBS2320 20 mg | MBS2320 40 mg
Number analyzed (Participants) | 62 | 62 | 63 | 61
percentage of patients | 48.4 | 49.2 | 42.4 | 57.7

2. Secondary Outcome: Safety and Tolerability of MBS2320
Description: Incidence of all grade adverse events
Time Frame: Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, a period of 12 weeks.
Arm/Group | Placebo | MBS2320 5 mg | MBS2320 20 mg | MBS2320 40 mg
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/63 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/63 | 2/61
Other Adverse Events (participants affected / at risk) | 4/62 | 16/62 | 8/63 | 13/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=62) | MBS2320 5 mg (N=62) | MBS2320 20 mg (N=63) | MBS2320 40 mg (N=61)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=62) | MBS2320 5 mg (N=62) | MBS2320 20 mg (N=63) | MBS2320 40 mg (N=61)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood bicarbonate decreased (Investigations) | 4 (4) | 4 (4) | 4 (4) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT05460832/Prot_SAP_000.pdf